CLINICAL TRIAL: NCT05582746
Title: Localized mHealth Approach to Boosting COVID-19 Testing and Vaccine Literacy, Access, and Uptake Among Women With Criminal Legal System Involvement
Brief Title: COVID-19 Testing and Vaccine Literacy for Women With Criminal Legal System Involvement
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jason E Glenn, PhD, Associate Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00148911; 5U01MD017415-02 (NIH)
Record Dates: First submitted 2022-10-05; First posted 2022-10-17 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 mHealth Intervention (Other): We are using a pre-post study design, given the low risk of the educational intervention and expected benefit.
  Interventions: Behavioral: Tri-City COVID Attitudes Study

INTERVENTIONS:
Behavioral: Tri-City COVID Attitudes Study — We propose a two-year study to rapidly assess (Aim 1), build and push (Aim 2), evaluate and disseminate (Aim 3) an mHealth intervention to boost COVID-19 testing and vaccine literacy, access, and uptake among women with CLSI in three cities

SUMMARY:
The objective of this research is to use a localized mHealth intervention to boost COVID-19 testing and vaccine literacy, access, and uptake among women with CLSI

DETAILED DESCRIPTION:
Based on our prior work with CLSI women, mHealth strategies are an excellent way to keep in touch and push just-in-time content. During the pandemic, we were forced to close field sites and stop any in-person follow-up visits. Even prior to the pandemic, telephone follow-up surveys were conducted with 60% of participants. Post-pandemic, we conducted 95% of those surveys over the phone, with the remaining over email or mail correspondence. Most participants use text messaging regularly and can access the Web on their phones. Our ongoing RCT (N=73 participants completed) of an mHealth intervention on women's health shows this modality is feasible for delivering information and engaging participants. Specifically, we found that 81% of women who initiate can complete the intervention. The average time for completion of one module, for example on sexually transmitted infections, took 19 minutes, whereas cervical cancer took 13 minutes to complete. We estimate the proposed module on COVID-19 testing and vaccine will take on average between 15 to 20 minutes to complete. This time for intervention completion, combined with text message information about any new COVID-19 mitigation news (e.g., boosters, vaccine for children, new testing recommendations, testing locations, etc.), should result in about 30-60 minutes of total formal engagement during the study.

What we propose will be brief, but targeted messaging intervention from verified sources, delivered in an adequate lay language and using spokespersons that are relatable and familiar, and can be trusted, has been proven effective in changing targeted behaviors.32,33 Our intervention design also draws on lessons learned from evidence-based interventions to improve vaccination uptake among adults, for example a meta-analysis conducted in 2021 on public response to health messages encouraging vaccination.34 Our mHealth intervention allows participants to attend to the information at their own pace, while ensuring that they are prompted to complete the module. To avoid unidirectionality and promote engagement, they will be able to use an asynchronous messaging component to ask questions and receive answers from the research team. There is no question that such an intervention is necessary for a population with likely low uptake of both testing and vaccination, especially when that population is not the explicit target of most public health messaging. To the critique of whether the intervention is sufficient, we don't know. We hypothesize that the intervention will be effective at boosting COVID-19 testing and vaccine literacy, access, and uptake, and the goal of this study is to test that hypothesis. One advantage of this approach is the ability for nimbleness, that is, being able to adapt in real-time to new information about the pandemic and being able to push that new information out to women using the proposed intervention platform. Another unique advantage is the scalability of such an intervention, and its ability to be made widely available to all CLSI women in the United States

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled in the Tri-City C.R.E.W. study (R01CA226838)

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Glenn, PHD, Principal Investigator — University of Kansas School of Medicine
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data generated through this application will be presented at scientific meetings annually, and in a timely manner, the final dataset will be published in peer-reviewed journals in the form of research articles. Efforts will be made to publish in journals open online to the public. De-identified data generated from this project, as well as data collection instruments will be shared publicly on the Coordination and Data Collection Center (CDCC) and the NIH RADx Data Hub, as well as on the Open Science Framework, a free, open-source research management and collaboration tool designed to help researchers document their project's lifecycle and archive materials. It is built and maintained by the nonprofit Center for Open Science. The final peer-reviewed journal manuscripts that arise from this NIH support will be submitted to the digital archive PubMed Central, per the NIH Public Access policy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: on-going
Access Criteria: access to the RAD-x DATA HUB via eRA account
URL: https://radx-hub.nih.gov/home

REFERENCES:
- [Background] Saloner B, Parish K, Ward JA, DiLaura G, Dolovich S. COVID-19 Cases and Deaths in Federal and State Prisons. JAMA. 2020 Aug 11;324(6):602-603. doi: 10.1001/jama.2020.12528. PMID 32639537
- [Background] Khorasani SB, Koutoujian PJ, Zubiago J, Guardado R, Siddiqi K, Wurcel AG. COVID-19 Vaccine Interest among Corrections Officers and People Who Are Incarcerated at Middlesex County Jail, Massachusetts. J Urban Health. 2021 Aug;98(4):459-463. doi: 10.1007/s11524-021-00545-y. Epub 2021 May 26. No abstract available. PMID 34041670
- [Background] Wickliffe J, Kelly PJ, Allison M, Emerson A, Ramaswamy M. Retention Strategies in Working With Justice-Involved Women. J Correct Health Care. 2019 Jul;25(3):231-237. doi: 10.1177/1078345819853310. Epub 2019 Jun 26. PMID 31242801
- [Background] Volpp KG, Cannuscio CC. Incentives for Immunity - Strategies for Increasing Covid-19 Vaccine Uptake. N Engl J Med. 2021 Jul 1;385(1):e1. doi: 10.1056/NEJMp2107719. Epub 2021 May 26. No abstract available. PMID 34038633
- [Background] Geana MV, Anderson S, Ramaswamy M. COVID-19 vaccine hesitancy among women leaving jails: A qualitative study. Public Health Nurs. 2021 Sep;38(5):892-896. doi: 10.1111/phn.12922. Epub 2021 May 11. PMID 33973268
- [Background] Ramaswamy M, Hemberg J, Faust A, Wickliffe J, Comfort M, Lorvick J, Cropsey K. Criminal Justice-Involved Women Navigate COVID-19: Notes From the Field. Health Educ Behav. 2020 Aug;47(4):544-548. doi: 10.1177/1090198120927304. Epub 2020 May 8. PMID 32380869
- [Background] Biasio LR, Bonaccorsi G, Lorini C, Pecorelli S. Assessing COVID-19 vaccine literacy: a preliminary online survey. Hum Vaccin Immunother. 2021 May 4;17(5):1304-1312. doi: 10.1080/21645515.2020.1829315. Epub 2020 Oct 29. PMID 33118868
- [Background] Bogart LM, Ojikutu BO, Tyagi K, Klein DJ, Mutchler MG, Dong L, Lawrence SJ, Thomas DR, Kellman S. COVID-19 Related Medical Mistrust, Health Impacts, and Potential Vaccine Hesitancy Among Black Americans Living With HIV. J Acquir Immune Defic Syndr. 2021 Feb 1;86(2):200-207. doi: 10.1097/QAI.0000000000002570. PMID 33196555
- [Background] Lipnicky A, Kelly PJ, Ramaswamy M. Facebook as a follow-up tool for women with criminal justice histories. Int J Prison Health. 2020 Apr 10;16(2):117-122. doi: 10.1108/IJPH-08-2019-0042. PMID 33634650
- [Background] Zhang Y, Fisk RJ. Barriers to vaccination for coronavirus disease 2019 (COVID-19) control: experience from the United States. Glob Health J. 2021 Mar;5(1):51-55. doi: 10.1016/j.glohj.2021.02.005. Epub 2021 Feb 9. PMID 33585053
- [Background] LaVeist TA, Nickerson KJ, Bowie JV. Attitudes about racism, medical mistrust, and satisfaction with care among African American and white cardiac patients. Med Care Res Rev. 2000;57 Suppl 1:146-61. doi: 10.1177/1077558700057001S07. PMID 11092161

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 mHealth Intervention: We are using a pre-post study design, given the low risk of the educational intervention and expected benefit. All participants received an mHealth intervention to boost COVID-19 testing and vaccine literacy, access, and uptake among women with CLSI in three cities.
Period: Baseline
Arm/Group | COVID-19 mHealth Intervention
Started | 295
Completed | 295
Not Completed | 0
Period: 1-month Follow-up
Arm/Group | COVID-19 mHealth Intervention
Started | 295
Completed | 265
Not Completed | 30
Period: 12-month Follow-up
Arm/Group | COVID-19 mHealth Intervention
Started | 265
Completed | 235
Not Completed | 30

BASELINE CHARACTERISTICS:
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There were n=10 (3.4%) missing for age.
  years
    number analyzed (Participants) | 285
    (all) | 45.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 256
  Unknown or Not Reported | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 172
  Race: White | 94
  Race: Other People of Color | 24
  Race: Unknown or not reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 295
Education [Count of Participants; unit: Participants]
  Less than High School | 59
  High School or higher | 227
  unknown or not reported | 9
Insurance [Count of Participants; unit: Participants]
  Yes | 244
  No | 36
  unknow or not reported | 15
Employment [Count of Participants; unit: Participants]
  Yes | 111
  No | 168
  Unknown or not reported | 16
City [Count of Participants; unit: Participants]
  Kansas City | 51
  Birmingham | 88
  Oakland | 156

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Testing and Vaccine Knowledge
Description: Nine multiple-choice items developed by study team and corresponding to intervention content, which regarding COVID-19 transmission, risk, mitigation, vaccine risk, and testing in a pandemic environment .
  The sum of scores on all 9 items has a possible total score ranges from 0 (minimum) to 9 (maximum), a higher score represents a higher level of COVID-19 testing and vaccine knowledge (i.e., better outcome).
Time Frame: Pre-Intervention assessment measured at baseline, Post-intervention assessment measured at 1-month and 12-month follow-ups.
Population: There is missing data due to no response, measures reported are reported before multiple imputation for missingness (i.e., only complete cases).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
score on a scale
  Pre-intervention assessment: number analyzed (Participants) | 287
  Pre-intervention assessment | 3.58 (1.36)
  1-month assessment: number analyzed (Participants) | 274
  1-month assessment | 3.98 (1.36)
  12-month assessment: number analyzed (Participants) | 243
  12-month assessment | 3.85 (1.39)

2. Primary Outcome: COVID-19 Mistrust Score
Description: General COVID-19 Mistrust Scale (PMID: 33196555) Adopted 4-items COVID-19 Mistrust Scale, which focus on public information advanced by the government and public health care providers.
  Each item was on 5-point Likert Scare range from 1 (strongly disagree) to 5 (strongly agree).
  A mean score of 4 items represent participants' mistrust level towards government and public health care providers, which ranges from 1 (minimum) to 5 (maximum).
  A higher score means a higher mistrust score (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
score on a scale
  Pre-intervention assessment: number analyzed (Participants) | 278
  Pre-intervention assessment | 3.25 (1.21)
  1-month assessment: number analyzed (Participants) | 269
  1-month assessment | 3.09 (1.16)
  12-month assessment: number analyzed (Participants) | 237
  12-month assessment | 3.21 (1.08)

3. Primary Outcome: COVID-19 Testing Accessibility - Ease of Access
Description: Self-reported perceived accessibility of COVID-19 testing. A 5-point Likert scale item ranges from 1 (strongly disagree) to 5 (strongly agree).
  A higher score represent participants' higher level of perceived accessibility (i.e., a better outcome).
Time Frame: as for outcome 1
Population: Pre-Intervention assessment measured at baseline, Post-intervention assessment measured at 1-month and 12-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
score on a scale
  Pre-Intervention assessment: number analyzed (Participants) | 287
  Pre-Intervention assessment | 4.36 (1.03)
  1-month: number analyzed (Participants) | 272
  1-month | 4.51 (0.89)
  12-month: number analyzed (Participants) | 240
  12-month | 4.49 (0.96)

4. Primary Outcome: COVID-19 Testing Accessibility - Confidence to Locate
Description: Self-reported confidence level of locating the place to get COVID-19 testing. A 5-point Likert scale item ranges from 1 (strongly disagree) to 5 (strongly agree).
  A higher score represent participants' higher level of confidence (i.e., a better outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
score on a scale
  Pre-Intervention assessment: number analyzed (Participants) | 287
  Pre-Intervention assessment | 4.42 (1.05)
  1-month assessment: number analyzed (Participants) | 269
  1-month assessment | 4.54 (0.95)
  12-month assessment: number analyzed (Participants) | 240
  12-month assessment | 4.49 (0.96)

5. Primary Outcome: COVID-19 Testing Accessibility - Free Access
Description: Percentage of participants' aware the government program that offers free tests through the mail.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
Participants
  Pre-Intervention assessment: number analyzed (Participants) | 283
  Pre-Intervention assessment | 209
  1-month assessment: number analyzed (Participants) | 267
  1-month assessment | 221
  12-month assessment: number analyzed (Participants) | 238
  12-month assessment | 195

6. Primary Outcome: Ever Had COVID-19 Testing
Description: Count number of participants who indicated they ever had COVID-19 testing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
Participants
  Pre-Intervention assessment: number analyzed (Participants) | 285
  Pre-Intervention assessment | 264
  1-month assessment: number analyzed (Participants) | 269
  1-month assessment | 253
  12-month assessment: number analyzed (Participants) | 239
  12-month assessment | 229

7. Primary Outcome: Ever Received COVID-19 Vaccine
Description: Count number of participants who indicated they ever had COVID-19 vaccine.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 mHealth Intervention
Number analyzed (Participants) | 295
Participants
  Pre-Intervention assessment: number analyzed (Participants) | 286
  Pre-Intervention assessment | 191
  1-month assessment: number analyzed (Participants) | 265
  1-month assessment | 182
  12-month assessment: number analyzed (Participants) | 231
  12-month assessment | 165

ADVERSE EVENTS:
Time Frame: 1 month, 12 month
Description: The expected adverse event risk is minimal as the intervention is an online educational module. Adverse events and Other adverse events were not monitored. The research team has dedicated members keep a record of any reported death at 1-month and 12-month follow-ups via non-systematic assessment.
Arm/Group | COVID-19 mHealth Intervention
All-Cause Mortality (participants affected / at risk) | 3/295
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT05582746/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT05582746/ICF_001.pdf